CLINICAL TRIAL: NCT00600340
Title: A Randomized Phase III 2-arm Trial of Paclitaxel Plus Bevacizumab vs. Capecitabine Plus Bevacizumab for the First-line Treatment of Human Epidermal Growth Factor Receptor 2 (HER2)-Negative Locally Recurrent or Metastatic Breast Cancer
Brief Title: 2-arm Trial of Paclitaxel Plus Bevacizumab vs. Capecitabine Plus Bevacizumab
Acronym: TURANDOT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Central European Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CECOG/BC1.3.005
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-10

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Paclitaxel; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A Bev+Pac (Active Comparator): Bevacizumab plus Paclitaxel
  Interventions: Biological: Bevacizumab and Paclitaxel
- B Bev+Cap (Active Comparator): Bevacizumab plus Capecitabine
  Interventions: Biological: Bevacizumab and Capecitabine

INTERVENTIONS:
Biological: Bevacizumab and Paclitaxel — A: Bevacizumab 10 mg/kg i.v., days 1 and 15, every 4 weeks Paclitaxel 90 mg/m2, days 1, 8 and 15, every 4 weeks
  Arms: A Bev+Pac
Biological: Bevacizumab and Capecitabine — B:Bevacizumab 15 mg/kg i.v., day 1, every 3 weeks Capecitabine twice-daily 1000 mg/m², day 1 to 14, every 3 weeks
  Arms: B Bev+Cap

SUMMARY:
First-line treatment of patients with locally recurrent or metastatic, HER2-negative breast cancer who have not received prior chemotherapy for locally recurrent or metastatic disease.

DETAILED DESCRIPTION:
Arm A:

Bevacizumab 10 mg/kg intravenous (i.v.), days 1 and 15, every 4 weeks

Paclitaxel 90 mg/m2, days 1, 8 and 15, every 4 weeks

Arm B:

Bevacizumab 15 mg/kg i.v., day 1, every 3 weeks

Capecitabine 1000 mg/m² twice-daily, days 1-14, every 3 weeks

In both arms treatment will be given until first disease progression (PD), unacceptable toxicity or withdrawal of patient consent.

For patients who stop chemotherapy for any reason before PD (e.g. toxicity) the other treatment should be given as monotherapy until PD.

ELIGIBILITY:
Inclusion Criteria

1. Written informed consent obtained prior to any study-specific procedure.
2. Age ≥18 years.
3. Able to comply with the protocol.
4. Histologically or cytologically confirmed, HER2-negative, adenocarcinoma of the breast with measurable or non-measurable locally recurrent or metastatic disease, who are candidates for chemotherapy. Locally recurrent disease must not be amenable to radiotherapy or resection with curative intent.
5. Eastern Cooperative Oncology Group (ECOG) performance Status (PS) of 0-2.
6. Life expectancy more than 12 weeks.
7. Prior (neo)adjuvant chemotherapy is allowed provided that the last dose of chemotherapy was more than 6 months prior to randomization. However, if (neo)adjuvant chemotherapy was:

   * Taxane-based, patients are eligible only if they received their last taxane more than 12 months prior to randomization.
   * Anthracycline-based, the maximum cumulative dose of prior anthracycline therapy must not exceed 360 mg/m2 for doxorubicin and 720 mg/m2 for epirubicin.
8. Prior adjuvant radiotherapy is allowed as part of the treatment of early breast cancer provided that last fraction of radiotherapy occurred at least 6 months prior to randomization. Radiotherapy administered solely for the relief of metastatic bone pain is allowed prior to study entry, providing that:

   * no more than 30% of marrow-bearing bone was irradiated
   * the last fraction of radiotherapy was administered ≥ 3 weeks prior to randomization.
9. Adequate left ventricular ejection function (LVEF) at baseline, defined as LVEF ≥ 50% by either echocardiogram or multigated acquisition scan (MUGA).
10. Adequate hematological function

    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    * Platelet count ≥ 100 x 109/L
    * Hemoglobin ≥ 9 g/dL (may be transfused to maintain or exceed this level).
11. Adequate liver function

    * Total bilirubin ≤ 1.25 x upper normal limit (ULN)
    * Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) < 2.5 x ULN in patients without liver metastases; < 5.0 x ULN in patients with liver metastases.
12. Adequate renal function

    * Serum creatinine ≤ 1.25 x ULN or calculated creatinine clearance ≥ 50 mL/min.
    * Urine dipstick for proteinuria < +2. Patients discovered to have ≥ +2 proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate ≤ 1g of protein in 24 hours
13. The use of full-dose oral or parenteral anticoagulants is permitted as long as the patient has been on a stable level of anticoagulation for at least two weeks at the time of randomization

    * Patients on heparin treatment should have a baseline activated partial thromboplastin time (aPTT) between 1.5 - 2.5 times ULN or patients value before starting heparin treatment
    * Patients on low molecular weight heparins (LMWH) should receive daily dose of 1.5 - 2 mg/kg (of enoxaparin) or appropriate doses of the correspondent anticoagulant, according to package insert
    * Patients on coumarin derivatives should have an international normalized ratio (INR) between 2.0 and 3.0 assessed at baseline in two consecutive measurements 1-4 days apart
    * Patients not receiving anticoagulant medication must have an INR ≤ 1.5 and aPTT ≤ 1.5 times ULN within 7 days prior to randomization

Exclusion Criteria

1. Previous chemotherapy for metastatic or locally recurrent breast cancer.
2. Concomitant hormonal therapy for locally recurrent or metastatic disease. Note: previous hormonal therapy is allowed for adjuvant, locally recurrent or metastatic breast cancer, but must have been discontinued at least 3 weeks prior to randomization.
3. Previous radiotherapy for the treatment of metastatic disease (unless given for the relief of metastatic bone pain and with the precautions mentioned above).
4. Other primary tumors within the last 5 years, except for adequately controlled limited basal cell carcinoma of the skin, or carcinoma in situ of the cervix.
5. Pre-existing peripheral neuropathy NCI CTCAE grade > 2 at randomization.
6. Evidence of spinal cord compression or current evidence of central nervous system (CNS) metastases (even if previously treated). If suspected, the patient should be scanned by CT or magnetic resonance imaging (MRI) within 28 days prior to randomization to rule out spinal / CNS metastases.
7. History or evidence upon physical/neurological examination of CNS disease unrelated to cancer, unless adequately treated with standard medical therapy (e.g. uncontrolled seizures).
8. Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to randomization, or anticipation of the need for major surgery during the course of the study treatment.
9. Minor surgical procedures, including insertion of an indwelling catheter, within 24 hours prior to randomization.
10. Current or recent (within 10 days of first dose of bevacizumab) use of aspirin (> 325 mg/day) or clopidogrel (> 75 mg/day).
11. Chronic daily treatment with corticosteroids (dose of > 10 mg/day methylprednisolone equivalent) (excluding inhaled steroids).
12. History or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding.
13. Uncontrolled hypertension (systolic > 150 mmHg and/or diastolic > 100 mmHg).
14. Clinically significant (i.e. active) cardiovascular disease, requiring medication during the study and might interfere with regularity of the study treatment, or not controlled by medication.
15. Non-healing wound, active peptic ulcer or bone fracture.
16. History of abdominal fistula, or any grade 4 non-gastrointestinal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months of randomization.
17. Active infection requiring i.v. antibiotics at randomization.
18. Pregnant or lactating females. Serum pregnancy test to be assessed within 7 days prior to study treatment start, or within 14 days with a confirmatory urine pregnancy test within 7 days prior to study treatment start.
19. Women of childbearing potential (< 2 years after the last menstruation) not using effective, non-hormonal means of contraception (intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly or surgically sterile) during the study and for a period of 6 months following the last administration of study drug.
20. Men who do not agree to use effective contraception during the study and for a period of 6 months following the last administration of study drug.
21. Current or recent (within 28 days of randomization) treatment with another investigational drug or participation in another investigational study
22. Clinically significant malabsorption syndrome or inability to take oral medication.
23. Psychiatric disability judged by the Investigator to be interfering with compliance for oral drug intake.
24. Requirement for concurrent use of the antiviral agent sorivudine or chemically related analogues, such as brivudine.
25. Evidence of any other disease, metabolic or psychological dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, or that may affect patient compliance with study routines, or places the patient at high risk from treatment related complications.
26. Known Dihydropyrimidine Dehydrogenase (DPD) deficiency or prior unanticipated severe reaction to fluoropyrimidine therapy (with or without documented DPD deficiency)
27. Known hypersensitivity to any of the study drugs (including 5-FU) or excipients. Hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies. History of hypersensitivity reactions with drugs formulated in Cremophor® EL (polyoxyethylated castor oil), or previous therapy with bevacizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2008-04; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph C Zielinski, MD, Principal Investigator — Dep. of Internal Medicin I, Oncology, Medical University of Vienna
Locations (55):
- Austria (8):
  - LKH Leoben, Leoben
  - Hospital Barmherzige Schwestern, Linz
  - AKH Linz, Dep. of Oncology, Linz
  - Hospital Elisabethinen Linz, Linz
  - Univ. Klinik, Medicine III, Salzburg
  - 2. Med. Abteilung - LKH-Steyr, Steyr
  - General Hospital, Medical University of Vienna, Vienna
  - Hospital Hietzing, Vienna
- Institute of Oncology Sarajevo, Sarajevo, Bosnia and Herzegovina
- Bulgaria (3):
  - Cancer Center Plovdiv, Plovdiv
  - University Hospital "Queen Joanna", Sofia
  - Interdistrict Oncology Dispensary, Varna
- Croatia (5):
  - Department for Oncology, GH Osijek, Osijek
  - General Hospital Pula, Pula
  - University Hospital Centre Rijeka, Rijeka
  - University Hospital for Tumors, Zagreb
  - University Hospital Rebro, Zagreb
- Czechia (4):
  - Krajska nemocnice Liberec, Liberec
  - Institut onkologie a rehablilitace na Plesi, Nová Ves pod Pleší
  - Fakultni nemocnice Olomouc, Olomouc
  - Charles University Prague, Dep of Oncology, Prague
- Hungary (4):
  - Semmelweis Univ. Radiology Clinic, Budapest
  - National Institute of Oncology, Budapest
  - Onkotherápiás Klinika,, Szeged
  - Markusovszky Teaching Hospital, Szombathely
- Israel (5):
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Assuta Medical Center, Tel Aviv
  - Tel Aviv Sourasky Medical Center, Div of Oncology, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
- Latvia (2):
  - P. Stradins University Hospital, Riga
  - Riga Eastern Hospital - the latvian Center of Oncology, Riga
- Poland (9):
  - Wojewodzkie Centrum Onkologii, Gdansk
  - Medical University of Gdansk, Gdansk
  - Klinika Onkologii CMuJ, Krakow
  - Lodz Oncology Center, Lodz
  - Centrum Medyczne Poradnia Onkologiczna, Rzeszów
  - Wojewodzki Szpital Specialistyczny, Siedlce
  - Szpital Wojewodzki im Sw. Lukasza, Tarnów
  - Memorial Cancer Center and Institute, Warsaw
  - Dolnoslaskie Centrum Onkologii, Wroclaw
- Romania (6):
  - Emergency University Bucharest Hospital, Bucharest
  - Institutul Oncologic Bucuresti, Bucharest
  - Cancer Institute "I. Chiricuta", Cluj-Napoca
  - University Hospital St. Spiridon Iasi, Iași
  - Clinical County Hospital Sibiu, Sibiu
  - Oncomed-Oncology Practice, Timișoara
- Serbia (4):
  - Institute for Oncology and Radiology, Belgrade
  - Clinical Hospital Center " Bezanijska Kosa", Belgrade
  - Institute of Oncology, Kamenitz
  - Clinic of Oncology, Niš
- Slovakia (4):
  - Nomocnica Sv. Alzbety, Narodny Onkologicky Ustav, Bratislava
  - National Cancer Institute, Bratislava
  - Oncology Institute, Department of Radiotherapy and Onclogy, Košice
  - POKO Porad, s.r.o, Poprad

REFERENCES:
- [Derived] Hoon SN, Lau PK, White AM, Bulsara MK, Banks PD, Redfern AD. Capecitabine for hormone receptor-positive versus hormone receptor-negative breast cancer. Cochrane Database Syst Rev. 2021 May 26;5(5):CD011220. doi: 10.1002/14651858.CD011220.pub2. PMID 34037241
- [Derived] Zielinski C, Lang I, Inbar M, Kahan Z, Greil R, Beslija S, Stemmer SM, Zvirbule Z, Steger GG, Melichar B, Pienkowski T, Sirbu D, Petruzelka L, Eniu A, Nisenbaum B, Dank M, Anghel R, Messinger D, Brodowicz T; TURANDOT investigators. Bevacizumab plus paclitaxel versus bevacizumab plus capecitabine as first-line treatment for HER2-negative metastatic breast cancer (TURANDOT): primary endpoint results of a randomised, open-label, non-inferiority, phase 3 trial. Lancet Oncol. 2016 Sep;17(9):1230-9. doi: 10.1016/S1470-2045(16)30154-1. Epub 2016 Aug 5. PMID 27501767
- [Derived] Brodowicz T, Lang I, Kahan Z, Greil R, Beslija S, Stemmer SM, Kaufman B, Petruzelka L, Eniu A, Anghel R, Koynov K, Vrbanec D, Pienkowski T, Melichar B, Spanik S, Ahlers S, Messinger D, Inbar MJ, Zielinski C. Selecting first-line bevacizumab-containing therapy for advanced breast cancer: TURANDOT risk factor analyses. Br J Cancer. 2014 Nov 25;111(11):2051-7. doi: 10.1038/bjc.2014.504. Epub 2014 Sep 30. PMID 25268370
- [Derived] Lang I, Brodowicz T, Ryvo L, Kahan Z, Greil R, Beslija S, Stemmer SM, Kaufman B, Zvirbule Z, Steger GG, Melichar B, Pienkowski T, Sirbu D, Messinger D, Zielinski C; Central European Cooperative Oncology Group. Bevacizumab plus paclitaxel versus bevacizumab plus capecitabine as first-line treatment for HER2-negative metastatic breast cancer: interim efficacy results of the randomised, open-label, non-inferiority, phase 3 TURANDOT trial. Lancet Oncol. 2013 Feb;14(2):125-33. doi: 10.1016/S1470-2045(12)70566-1. Epub 2013 Jan 10. PMID 23312888

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab Plus Paclitaxel: Bevacizumab 10 mg/kg i.v., days 1 and 15, every 4 weeks, Paclitaxel 90 mg/m2, days 1, 8 and 15, every 4 weeks
- Bevacizumab Plus Capecitabine: Bevacizumab 15 mg/kg i.v., day 1, every 3 weeks, Capecitabine twice-daily 1000 mg/m², day 1 to 14, every 3 weeks
Period: Overall Study
Arm/Group | Bevacizumab Plus Paclitaxel | Bevacizumab Plus Capecitabine
Started | 285 | 279
Completed | 285 | 279
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat Population (ITT)
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab Plus Paclitaxel | Bevacizumab Plus Capecitabine | Total
Number analyzed (Participants) | 285 | 279 | 564
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 218 | 201 | 419
  >=65 years | 67 | 78 | 145
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [49 to 64] | 59 [48 to 65] | 59 [49 to 65]
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (10.98) | 56.6 (11.67) | 56.6 (11.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 284 | 275 | 559
  Male | 1 | 4 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/ White | 283 | 278 | 561
  Black | 1 | 0 | 1
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Austria | 38 | 37 | 75
  Latvia | 15 | 12 | 27
  Romania | 20 | 22 | 42
  Hungary | 82 | 80 | 162
  Czechia | 18 | 19 | 37
  Poland | 19 | 17 | 36
  Slovakia | 6 | 9 | 15
  Israel | 54 | 51 | 105
  Bulgaria | 7 | 6 | 13
  Serbia | 6 | 8 | 14
  Bosnia and Herzegovina | 13 | 13 | 26
  Croatia | 7 | 5 | 12
Menopausal status [Count of Participants; unit: Participants]
  Pre-menopausal | 52 | 52 | 104
  Post-menopausal | 232 | 223 | 455
  Male patients | 1 | 4 | 5
Eastern Cooperative Oncology Group Performance Status (ECOG PS) [Count of Participants; unit: Participants] — 0 - Asymptomatic, 1 - Symptomatic but completely ambulatory, 2 - Symptomatic, <50% in bed during the day, 3 - Symptomatic, >50% in bed, but not bedbound, 4 - Bedbound, 5 - Death
  Participants
    0 | 193 | 179 | 372
    1 | 75 | 91 | 166
    2 | 16 | 7 | 23
    Missing | 1 | 2 | 3
Estrogen receptor (ER) [Count of Participants; unit: Participants]
  Positive | 215 | 201 | 416
  Negative | 68 | 77 | 145
  Unknown | 2 | 1 | 3
Progesterone Receptor (PgR) [Count of Participants; unit: Participants]
  Positive | 167 | 168 | 335
  Negative | 118 | 109 | 227
  Unknown | 0 | 2 | 2
Estrogen and progesterone receptor [Count of Participants; unit: Participants]
  ER and PgR negative | 63 | 67 | 130
  ER or PgR positive | 221 | 212 | 433
  ER and PR unknown or negative | 1 | 0 | 1
Electrocardiogram (ECG) result [Count of Participants; unit: Participants]
  Normal | 243 | 246 | 489
  Abnormal | 39 | 30 | 69
  Not performed | 3 | 3 | 6
Method for brain imaging [Count of Participants; unit: Participants] — No brain CT or MRI was required if the patient did not show signs/symptoms of central nervous system (CNS) involvement or other unexplained neurological symptoms.
  Participants
    CT | 18 | 19 | 37
    MRI | 3 | 2 | 5
    No brain CT/MRI | 264 | 258 | 522
Result of brain CT/MRI [Count of Participants; unit: Participants] — No brain CT or MRI was required if the patient did not show signs/symptoms suggestive of CNS involvement or other unexplained neurological symptoms.
  Participants
    No metastasis | 21 | 21 | 42
    No brain CT/MRI | 264 | 258 | 522
Stage at primary diagnosis: Primary tumor (T) [Count of Participants; unit: Participants] — Tis - Ductal carcinoma in situ, TX - Primary Tumor cannot be assessed, T1 - Tumor ≤ 20 mm in greatest dimension, T2 - Tumor > 20 mm but ≤ 50 mm in greatest dimension, T3 - Tumor > 50 mm in greatest dimension, T4 - Tumor of any size with direct extension to chest wall and/or to skin (ulceration or macroscopic nodules).
  Participants
    Tis | 1 | 2 | 3
    T1 | 66 | 72 | 138
    T2 | 130 | 118 | 248
    T3 | 26 | 32 | 58
    T4 | 45 | 38 | 83
    TX | 16 | 16 | 32
    Missing | 1 | 1 | 2
Stage at primary diagnosis: Regional lymph nodes (N) [Count of Participants; unit: Participants] — Nx - Regional lymph nodes cannot be assessed, N0 - No regional lymph node metastases, N1 - Metastases to movable ipsilateral level I, II axillary lymph nodes, N2 - Metastases in ipsilateral level I, II axillary lymph nodes that are clinically fixed or matted; or in clinically detected ipsilateral internal mammary nodes in absence of clinically evident axillary lymph node metastases, N3 - Metastases in ipsilateral infraclavicular (level III axillary) lymph nodes with or without level I, II axillary lymph node involvement.
  Participants
    N0 | 78 | 62 | 140
    N1 | 97 | 116 | 213
    N2 | 55 | 51 | 106
    N3 | 26 | 22 | 48
    NX | 28 | 27 | 55
    Missing | 1 | 1 | 2
Stage at primary diagnosis: Distant metastasis (M) [Count of Participants; unit: Participants] — M0 - No clinical or radiographic evidence of distant metastases, M1 - Distant metastases detected, Mx - Metastases cannot be assessed.
  Participants
    M0 | 222 | 219 | 441
    M1 | 62 | 59 | 121
    Missing | 1 | 1 | 2
Current stage of locally recurrent/ metastatic tumor [Count of Participants; unit: Participants]
  Locally recurrent breast cancer | 2 | 0 | 2
  Metastatic breast cancer | 282 | 279 | 561
  Missing | 1 | 0 | 1
Disease free interval after therapy of primary breast cancer [Count of Participants; unit: Participants]
  Yes | 214 | 215 | 429
  No | 71 | 64 | 135
Disease free interval [Count of Participants; unit: Participants] — Disease free interval set to 0 months (No DFI), if the patient did not receive previous therapy for primary breast cancer or if the patient was not disease free after previous therapy of primary breast cancer
  Participants
    No DFI | 71 | 64 | 135
    DFI <=12 months | 14 | 10 | 24
    DFI >12 and <=24 months | 52 | 34 | 86
    DFI >24 months | 148 | 171 | 319
Metastatic lesions [Count of Participants; unit: Participants] — All sites with at least one metastatic lesion. Patients can have multiple sites with metastatic lesions.
  Participants
    At least one metastatic lesion | 282 | 279 | 561
    Bone | 158 | 151 | 309
    Lung | 112 | 122 | 234
    Liver | 113 | 126 | 239
    Skin | 13 | 9 | 22
    Soft tissue | 69 | 63 | 132
    Lymph nodes | 146 | 171 | 317
    Other | 19 | 25 | 44
    Lung and / or liver | 185 | 203 | 388
    Soft tissue and/or bone only | 41 | 23 | 64
Imaging methods [Count of Participants; unit: Participants]
  CT | 270 | 261 | 531
  MRI | 8 | 12 | 20
  X-ray | 7 | 6 | 13
Target and non-target lesions [Count of Participants; unit: Participants]
  Target lesions only | 34 | 22 | 56
  Non-target lesions only | 65 | 49 | 114
  Both | 185 | 208 | 393
  None | 1 | 0 | 1
Number of target lesions [Count of Participants; unit: Participants]
  0 lesions | 66 | 49 | 115
  1 lesions | 48 | 49 | 97
  2 lesions | 41 | 49 | 90
  3 lesions | 47 | 39 | 86
  4-5 lesions | 44 | 57 | 101
  >= 6 lesions | 39 | 36 | 75
Sum of longest diameter of target lesion [Count of Participants; unit: Participants]
  No lesions | 66 | 49 | 115
  1-5 cm | 86 | 83 | 169
  >5-10 cm | 64 | 77 | 141
  >10 cm | 69 | 70 | 139
Number of organs with metastases [Count of Participants; unit: Participants]
  >= 3 | 105 | 124 | 229
  < 3 | 180 | 155 | 335
Previous hormonal therapy [Count of Participants; unit: Participants] — LR/MBC = for locally recurrent / metastatic breast cancer
  Participants
    Neoadjuvant/adjuvant only | 113 | 112 | 225
    LR/MBC only | 25 | 33 | 58
    Both | 37 | 25 | 62
    Other | 0 | 1 | 1
    None | 110 | 108 | 218
Neoadjuvant/ adjuvant hormonal therapy only [Count of Participants; unit: Participants] — Population: Only participants with neoadjuvant/adjuvant hormonal therapy included. Multiple answers per patient possible.
  Participants
    Anti-estrogens: number analyzed (Participants) | 113 | 112 | 225
    Anti-estrogens | 87 | 89 | 176
    Aromatase inhibitors: number analyzed (Participants) | 113 | 112 | 225
    Aromatase inhibitors | 56 | 56 | 112
    LR-RH analogues: number analyzed (Participants) | 113 | 112 | 225
    LR-RH analogues | 12 | 15 | 27
    Progesterone: number analyzed (Participants) | 113 | 112 | 225
    Progesterone | 0 | 1 | 1
    Other: number analyzed (Participants) | 113 | 112 | 225
    Other | 0 | 1 | 1
Hormonal therapy for LR/MBC only [Count of Participants; unit: Participants] — Population: Only participants with hormonal therapy for LR/ MBC included. Multiple answers per patient possible.
  Participants
    Anti-estrogens: number analyzed (Participants) | 25 | 33 | 58
    Anti-estrogens | 18 | 29 | 47
    Aromatase inhibitors: number analyzed (Participants) | 25 | 33 | 58
    Aromatase inhibitors | 17 | 23 | 40
    LH-RH analogues: number analyzed (Participants) | 25 | 33 | 58
    LH-RH analogues | 1 | 4 | 5
Previous neoadjuvant chemotherapy [Count of Participants; unit: Participants]
  Anthracycline and taxane | 16 | 11 | 27
  Anthracycline, no taxane | 41 | 33 | 74
  Taxane, no anthracycline | 5 | 5 | 10
  No anthracycline, no taxane, other | 2 | 3 | 5
  None | 221 | 227 | 448
Previous adjuvant chemotherapy [Count of Participants; unit: Participants]
  Anthracycline and taxane | 21 | 25 | 46
  Anthracycline, no taxane | 83 | 89 | 172
  Taxane, no anthracycline | 16 | 12 | 28
  No anthracycline, no taxane, other | 30 | 25 | 55
  None | 135 | 128 | 263
Previous neoadjuvant/adjuvant chemotherapy [Count of Participants; unit: Participants] — Patients for whom their neoadjuvant and adjuvant chemotherapy differed are counted in both the pertinent categories.
  Participants
    Anthracycline and taxane | 37 | 35 | 72
    Anthracycline, no taxane | 110 | 112 | 222
    Taxane, no anthracycline | 21 | 16 | 37
    No anthracycline, no taxane, other | 32 | 28 | 60
    None | 105 | 103 | 208
Previous neoadjuvant/adjuvant chemotherapy medications [Count of Participants; unit: Participants] — Patients who received both anthracycline and taxane in an adjuvant or neoadjuvant chemotherapy are counted in both categories.
  Participants
    Anthracycline | 145 | 144 | 289
    Taxane | 57 | 50 | 107
    No anthracycline, no taxane, other | 26 | 26 | 52
    None | 105 | 103 | 208
Previous radiotherapy [Count of Participants; unit: Participants] — Multiple answers per patient possible. In case of multiple treatments in the same category, the patient is counted only once in that category. Population: Restricted to patients with previous radiotherapy.
  Participants
    Neoadjuvant: number analyzed (Participants) | 191 | 194 | 385
    Neoadjuvant | 8 | 9 | 17
    Adjuvant: number analyzed (Participants) | 191 | 194 | 385
    Adjuvant | 167 | 171 | 338
    For relief of metastatic bone pain: number analyzed (Participants) | 191 | 194 | 385
    For relief of metastatic bone pain | 32 | 44 | 76
Previous surgery [Count of Participants; unit: Participants] — Multiple answers per patient possible. In case of multiple treatments in the same category, the patient is counted only once in that category. Population: Restricted to patients with previous surgery.
  Participants
    Total mastectomy: number analyzed (Participants) | 241 | 239 | 480
    Total mastectomy | 131 | 135 | 266
    Breast conserving surgery: number analyzed (Participants) | 241 | 239 | 480
    Breast conserving surgery | 111 | 99 | 210
    Biopsy/Aspiration: number analyzed (Participants) | 241 | 239 | 480
    Biopsy/Aspiration | 54 | 48 | 102
    Other: number analyzed (Participants) | 241 | 239 | 480
    Other | 35 | 29 | 64
Height [Mean (Standard Deviation); unit: cm] | 162 (6.60) | 162.3 (6.48) | 162.2 (6.54)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m²] | 1.76 (0.1834) | 1.773 (0.1688) | 1.767 (0.1763)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 127.9 (12.91) | 128.7 (13.85) | 128.3 (13.38)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 78.1 (8.23) | 77.9 (9.34) | 78.0 (8.79)
Heart rate [Mean (Standard Deviation); unit: bpm] | 79.7 (11.27) | 79.1 (11.41) | 79.4 (11.33)
Body temperature [Mean (Standard Deviation); unit: °C] | 36.55 (0.265) | 36.47 (0.305) | 36.51 (0.288)
Left Ventricular Ejection Fraction (LVEF) [Mean (Standard Deviation); unit: percentage of ejected blood] | 63.4 (5.32) | 62.6 (6.26) | 63.0 (5.81)
Time since diagnosis of adenocarcinoma [Mean (Standard Deviation); unit: months] — Histologically or cytologically confirmed adenocarcinoma.
  months | 55.2 (56.46) | 58.9 (55.09) | 57.0 (55.77)
Time since diagnosis of LR or MT [Mean (Standard Deviation); unit: months] — LR or MT = Locally recurrent or metastatic tumor.
  months | 5.7 (14.77) | 7.6 (19.11) | 6.7 (17.07)
Disease free interval [Mean (Standard Deviation); unit: months] — Disease free interval was set to 0 months (No DFI) if the patient did not receive previous therapy for primary breast cancer or the patient was not disease free after previous therapy for primary breast cancer.
  months | 43.6 (48.84) | 48.0 (48.53) | 45.8 (48.70)
Number of target lesions [Mean (Standard Deviation); unit: number of lesions] | 2.7 (2.52) | 2.8 (2.42) | 2.7 (2.47)
Sum of longest diameter of target lesions [Mean (Standard Deviation); unit: cm] | 6.758 (7.4372) | 6.872 (6.6679) | 6.815 (7.0610)
Weight [Mean (Standard Deviation); unit: kg] | 71.97 (15.679) | 72.90 (14.350) | 72.43 (15.030)

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (PP Population)
Description: Overall survival (OS) defined as time from randomization to date of death from any cause. Patients without recorded death were censored at the date the patient was last known to be alive. OS was analyzed at two looks, one interim look and the final analysis. Due to group sequential testing, the overall significance level alpha = 0.025 was spent on both looks according to Lan-DeMets spending method with O'Brien-Fleming-type boundaries. Alpha spent at Interim after 47% of information was 0.0010. Alpha spent at final analysis after 99% of information was 0.0250.
Time Frame: Time from the date of randomization to the date of death or date last known to be alive, assessed up to approximately 6 years
Population: Per Protocol Population (PP)
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bevacizumab Plus Paclitaxel: Bevacizumab 10 mg/kg intravenous (i.v.), days 1 and 15, every 4 weeks, Paclitaxel 90 mg/m2, days 1, 8 and 15, every 4 weeks
- Bevacizumab Plus Capecitabine: Bevacizumab 15 mg/kg i.v., day 1, every 3 weeks, Capecitabine 1000 mg/m² twice-daily, days 1-14, every 3 weeks
Arm/Group | Bevacizumab Plus Paclitaxel | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 266 | 265
months | 30.2 [25.6 to 32.6] | 26.1 [22.3 to 29.0]
Statistical Analysis 1: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; HR of Bevacizumab plus Capecitabine vs. Bevacizumab plus Paclitaxel for OS (interim, stratified); Test type: Non-Inferiority — Null hypothesis: Hazard Ratio (HR) >= 1.33 Based on Cox proportional hazards model adjusted by stratification factors at randomization: 1. estrogen and/or progesterone status (positive vs. other) 2. country 3. menopausal status (premenopausal or male <=50 years of age vs. postmenopausal or male >50 years of age); p = 0.1983, Regression, Cox — Based on approach using repeated confidence intervals, with one-sided 97.5% repeated confidence intervals; Hazard Ratio (HR) = 1.042, 97.5% CI 1-sided [upper limit 1.689] — HR is the hazard rate of Bevacizumab plus Capecitabine divided by hazard rate of Bevacizumab plus Paclitaxel
Statistical Analysis 2: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; HR of Bevacizumab Plus Capecitabine vs. Bevacizumab plus Paclitaxel for OS (final, stratified); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0070, Regression, Cox — Based on approach using repeated confidence intervals, with one-sided 97.5% repeated confidence intervals. Non-inferiority margin was a HR of 1.33; Hazard Ratio (HR) = 1.018, 97.5% CI 1-sided [upper limit 1.261] — HR is the hazard rate of Bevacizumab Plus Capecitabine divided by hazard rate of Bevacizumab plus Paclitaxel
Statistical Analysis 3: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; HR of Bevacizumab Plus Capecitabine vs. Bevacizumab plus Paclitaxel for OS (interim, unstratified); Test type: Non-Inferiority — Null hypothesis: Hazard Ratio (HR) >= 1.33 Based on Cox proportional hazards model; p = 0.2024, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 1.058, 97.5% CI 1-sided [upper limit 1.674] — HR is the hazard rate of Bevacizumab Plus Capecitabine divided by hazard rate of Bevacizumab plus Paclitaxel
Statistical Analysis 4: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; HR of Bevacizumab Plus Capecitabine vs. Bevacizumab plus Paclitaxel for OS (final, unstratified); Test type: Non-Inferiority — Null hypothesis: Hazard Ratio (HR) >= 1.33 Based on Cox proportional hazards model; p = 0.0612, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Hazard Ratio (HR) = 1.134, 97.5% CI 1-sided [upper limit 1.386] — HR is the hazard rate of Bevacizumab Plus Capecitabine divided by hazard rate of Bevacizumab plus Paclitaxel

2. Primary Outcome: Overall Survival (ITT Population)
Description: Overall survival (OS) defined as time from randomization to date of death from any cause. Patients without recorded death were censored at the date the patient was last known to be alive. OS was analyzed at two looks, one interim look and the final analysis. Due to group sequential testing, the overall significance level alpha = 0.025 was spent on both looks according to Lan-DeMets spending method with O'Brien-Fleming-type boundaries. Alpha spent at Interim after 50% of information was 0.0014. Alpha spent at final analysis after 99% of information was 0.0250.
Time Frame: as for outcome 1
Population: Intent-to-Treat Population (ITT)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab Plus Paclitaxel | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 285 | 279
months | 29.5 [25.3 to 32.4] | 26.0 [22.3 to 29.0]
Statistical Analysis 1: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; HR of Bevacizumab Plus Capecitabine vs. Bevacizumab plus Paclitaxel for OS (interim, stratified); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.1534, Regression, Cox — Based on approach using repeated confidence intervals, with one-sided 97.5% repeated confidence intervals; Hazard Ratio (HR) = 1.027, 97.5% CI 1-sided [upper limit 1.606] — HR is the hazard rate of Bevacizumab Plus Capecitabine divided by hazard rate of Bevacizumab plus Paclitaxel
Statistical Analysis 2: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; HR of Bevacizumab Plus Capecitabine vs. Bevacizumab plus Paclitaxel for OS (final, stratified); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0085, Regression, Cox — Based on approach using repeated confidence intervals, with one-sided 97.5% repeated confidence intervals; Hazard Ratio (HR) = 1.035, 97.5% CI 1-sided [upper limit 1.273] — HR is the hazard rate of Bevacizumab Plus Capecitabine divided by hazard rate of Bevacizumab plus Paclitaxel
Statistical Analysis 3: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; HR of Bevacizumab Plus Capecitabine vs. Bevacizumab plus Paclitaxel for OS (interim, unstratified); Test type: Non-Inferiority — Null hypothesis: Hazard Ratio (HR) >= 1.33 Based on Cox proportional hazards model; p = 0.1778, Regression, Cox — Based on approach using repeated confidence intervals, with one-sided 97.5% repeated confidence intervals; Hazard Ratio (HR) = 1.058, 97.5% CI 1-sided [upper limit 1.623] — HR is the hazard rate of Bevacizumab Plus Capecitabine divided by hazard rate of Bevacizumab plus Paclitaxel
Statistical Analysis 4: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; HR of Bevacizumab Plus Capecitabine vs. Bevacizumab plus Paclitaxel for OS (final, unstratified); Test type: Non-Inferiority — Null hypothesis: Hazard Ratio (HR) >= 1.33 Based on Cox proportional hazards model; p = 0.049, Regression, Cox — Based on approach using repeated confidence intervals, with one-sided 97.5% repeated confidence intervals; Hazard Ratio (HR) = 1.126, 97.5% CI 1-sided [upper limit 1.37] — HR is the hazard rate of Bevacizumab Plus Capecitabine divided by hazard rate of Bevacizumab plus Paclitaxel

3. Secondary Outcome: Observation Time (ITT Population)
Description: Median observation time estimated with reverse Kaplan-Meier methods. Observation time (in months) is defined as time from randomization to the day the patient was last confirmed to be alive. In case of patient deaths the time was censored at the day of death.
Time Frame: Up to approximately 6 years
Population: Intention-to-Treat population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab Plus Paclitaxel | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 285 | 279
months | 54.3 [53.1 to 57.5] | 55.7 [53.7 to 58.1]

4. Secondary Outcome: Best Overall Response (ITT Population)
Description: The best overall response according to the RECIST criteria is the best response recorded from the start of the treatment until disease progression/recurrence or within 28 days of last intake of study medication in the Study Treatment Phase
Time Frame: Up to disease progression or up to 28 days after last intake of study medication, assessed up to approximately 5 years.
Population: Intent-to-Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab Plus Paclitaxel | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 285 | 279
Participants
  Complete response | 10 | 2
  Partial response | 115 | 74
  Stable disease | 127 | 138
  Progressive disease | 18 | 47
  Not evaluable | 15 | 18

5. Secondary Outcome: Best Overall Response (PP Population)
Description: as for outcome 4
Time Frame: Up to disease progression or up to 28 days after last intake of study medication, assessed up to approximately 5 years.
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab Plus Paclitaxel | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 266 | 265
Participants
  Complete response | 10 | 2
  Partial response | 111 | 72
  Stable disease | 117 | 130
  Progressive disease | 17 | 45
  Not evaluable | 11 | 16

6. Secondary Outcome: Unconfirmed Best Overall Response (ITT Population)
Description: The best overall response according to the RECIST criteria is the best response recorded from the start of the treatment until disease progression/recurrence or within 28 days of last intake of study medication in the Study Treatment Phase. Complete and partial response in this summary did not require a confirmation by a second tumor assessment.
Time Frame: Up to disease progression or up to 28 days after last intake of study medication, assessed up to approximately 5 years.
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab Plus Paclitaxel | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 285 | 279
Participants
  Complete response | 16 | 4
  Partial response | 147 | 101
  Stable disease | 89 | 109
  Progressive disease | 18 | 47
  Not evaluable | 15 | 18

7. Secondary Outcome: Unconfirmed Best Overall Response (PP Population)
Description: as for outcome 6
Time Frame: Up to disease progression or up to 28 days after last intake of study medication, assessed up to approximately 5 years.
Population: PP population
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab Plus Paclitaxel | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 266 | 265
Participants
  Complete response | 16 | 4
  Partial response | 141 | 96
  Stable disease | 81 | 104
  Progressive disease | 17 | 45
  Not evaluable | 11 | 16

8. Secondary Outcome: Objective Response Rate and Disease Control Rate (ITT Population)
Description: Objective response rate (ORR) is defined as the proportion of patients with complete response or partial response. Disease control rate (DCR) is defined as the proportion of patients with complete response, partial response and stable disease. The best overall response according to the RECIST criteria is the best response recorded from the start of the treatment until disease progression/recurrence or within 28 days of last intake of study medication in the Study Treatment Phase
Time Frame: Up to disease progression or up to 28 days after last intake of study medication, assessed up to approximately 5 years.
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab Plus Paclitaxel | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 285 | 279
Participants
  Objective response | 125 | 76
  Disease control | 252 | 214
Statistical Analysis 1: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; Odds Ratio (OR) of objective response and Cochran-Mantel-Haenszel (CMH) test (stratified); Test type: Superiority — OR is the odds for objective response of Bevacizumab Plus Capecitabine divided by the odds for objective response of Bevacizumab plus Paclitaxel; p < 0.0001, Cochran-Mantel-Haenszel — Test adjusted by stratification factors at randomization: 1. estrogen and/or progesterone status (positive vs. other) 2. country 3. menopausal status (premenopausal or male <=50 years of age vs. postmenopausal or male >50 years of age; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.33 to 0.67] — OR is the odds for objective response of Bevacizumab Plus Capecitabine divided by the odds for objective response of Bevacizumab plus Paclitaxel
Statistical Analysis 2: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; Difference in ORR in Bevacizumab Plus Capecitabine vs. Bevacizumab plus Paclitaxel; Test type: Superiority; Risk Difference (RD) = -17, 95% CI 2-sided [-24 to -9] — Difference calculated as ORR in Bevacizumab Plus Capecitabine minus ORR in Bevacizumab plus Paclitaxel, units in percent
Statistical Analysis 3: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; OR of disease control and CMH test (stratified); Test type: Superiority — OR is the odds for disease control of Bevacizumab Plus Capecitabine divided by the odds for disease control of Bevacizumab plus Paclitaxel; p = 0.0006, Cochran-Mantel-Haenszel — [p-value comment as in outcome 8, analysis 1]; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.27 to 0.70] — OR is the odds for disease control of Bevacizumab Plus Capecitabine divided by the odds for disease control of Bevacizumab plus Paclitaxel
Statistical Analysis 4: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; Difference in DCR in Bevacizumab Plus Capecitabine vs. Bevacizumab plus Paclitaxel; Test type: Superiority; Risk Difference (RD) = -12, 95% CI 2-sided [-18 to -6] — Difference calculated as the DCR in Bevacizumab Plus Capecitabine minus ORR in Bevacizumab plus Paclitaxel, units in percent

9. Secondary Outcome: Objective Response Rate and Disease Control Rate (PP Population)
Description: as for outcome 8
Time Frame: Up to disease progression or up to 28 days after last intake of study medication, assessed up to approximately 5 years.
Population: PP population
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab Plus Paclitaxel | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 266 | 265
Participants
  Objective response | 121 | 74
  Disease control | 238 | 204
Statistical Analysis 1: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; OR of objective response and CMH test (stratified); Test type: Superiority — [test comment as in outcome 8, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 8, analysis 1]; Odds Ratio (OR) = 0.45, 95% CI 2-sided [0.31 to 0.65] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; Difference in ORR in Bevacizumab Plus Capecitabine vs. Bevacizumab plus Paclitaxel; Test type: Superiority; Risk Difference (RD) = -18, 95% CI 2-sided [-26 to -10] — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 3: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; OR of disease control and CMH test (stratified); Test type: Superiority — [test comment as in outcome 8, analysis 3]; p = 0.0003, Cochran-Mantel-Haenszel — [p-value comment as in outcome 8, analysis 1]; Odds Ratio (OR) = 0.39, 95% CI 2-sided [0.24 to 0.65] — [estimate comment as in outcome 8, analysis 3]
Statistical Analysis 4: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; Difference in DCR in Bevacizumab Plus Capecitabine vs. Bevacizumab plus Paclitaxel; Test type: Superiority; Risk Difference (RD) = -12, 95% CI 2-sided [-19 to -6] — [estimate comment as in outcome 8, analysis 4]

10. Secondary Outcome: Unconfirmed Objective Response Rate and Disease Control Rate (ITT Population)
Description: Objective response rate (ORR) is defined as the proportion of patients with complete response or partial response. Disease control rate (DCR) is defined as the proportion of patients with complete response, partial response and stable disease. The best overall response according to the RECIST criteria is the best response recorded from the start of the treatment until disease progression/recurrence or within 28 days of last intake of study medication in the Study Treatment Phase. Complete and partial response in this summary did not require a confirmation by a second tumor assessment.
Time Frame: Up to disease progression or up to 28 days after last intake of study medication, assessed up to approximately 5 years.
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab Plus Paclitaxel | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 285 | 279
Participants
  Objective response | 163 | 105
  Disease control | 252 | 214
Statistical Analysis 1: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; OR of objective response and CMH test (stratified); Test type: Superiority — [test comment as in outcome 8, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 8, analysis 1]; Odds Ratio (OR) = 0.44, 95% CI 2-sided [0.31 to 0.63] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; Difference in ORR in Bevacizumab Plus Capecitabine vs. Bevacizumab plus Paclitaxel; Test type: Superiority; Risk Difference (RD) = -20, 95% CI 2-sided [-28 to -11] — [estimate comment as in outcome 8, analysis 2]
Statistical Analysis 3: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; OR of disease control and CMH test (stratified); Test type: Superiority; p = 0.0006, Cochran-Mantel-Haenszel — [p-value comment as in outcome 8, analysis 1]; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.27 to 0.70] — [estimate comment as in outcome 8, analysis 3]
Statistical Analysis 4: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; Difference in DCR in Bevacizumab Plus Capecitabine vs. Bevacizumab plus Paclitaxel; Test type: Superiority; Risk Difference (RD) = -12, 95% CI 2-sided [-18 to -6] — Difference calculated as DCR in Bevacizumab Plus Capecitabine minus DCR in Bevacizumab plus Paclitaxel, units in percent

11. Secondary Outcome: Unconfirmed Objective Response Rate and Disease Control Rate (PP Population)
Description: as for outcome 10
Time Frame: Up to disease progression or up to 28 days after last intake of study medication, assessed up to approximately 5 years.
Population: PP population
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab Plus Paclitaxel | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 266 | 265
Participants
  Objective response | 157 | 100
  Disease control | 238 | 204
Statistical Analysis 1: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; OR of objective response and CMH test (stratified); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 8, analysis 1]; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.29 to 0.60] — [estimate comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; Difference in ORR in Bevacizumab Plus Capecitabine vs. Bevacizumab plus Paclitaxel; Test type: Superiority; Risk Difference (RD) = -21, 95% CI 2-sided [-30 to -13] — Difference calculated as ORR in Bevacizumab Plus Capecitabine minus ORR in Bevacizumab plus Paclitaxel, unit in percent
Statistical Analysis 3: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; OR of disease control and CMH test (stratified); Test type: Superiority — [test comment as in outcome 8, analysis 3]; p = 0.0003, Cochran-Mantel-Haenszel — [p-value comment as in outcome 8, analysis 1]; Odds Ratio (OR) = 0.39, 95% CI 2-sided [0.24 to 0.65] — [estimate comment as in outcome 8, analysis 3]
Statistical Analysis 4: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; Difference in DCR in Bevacizumab Plus Capecitabine vs. Bevacizumab plus Paclitaxel; Test type: Superiority; Risk Difference (RD) = -12, 95% CI 2-sided [-19 to -6] — Difference calculated as DCR in Bevacizumab Plus Capecitabine minus DCR in Bevacizumab plus Paclitaxel, unit in percent

12. Secondary Outcome: Progression Free Survival (ITT Population)
Description: Progression Free Survival (PFS) is defined as time from randomization to date of documented progression or date of death due to any cause, whichever occurred first. Patients without recorded progression or death were censored at the last date they were known to have not progressed. Patients who were randomized and had no post-baseline tumor assessment were censored on the day of randomization. Median PFS, associated stratified Hazard Ratio (HR).
Time Frame: Time from the date of randomization to disease progression, death or censoring (whichever occurred first), assessed up to approximately 5 years.
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab Plus Paclitaxel | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 285 | 279
months | 10.9 [10.3 to 12.9] | 8.1 [6.8 to 8.9]
Statistical Analysis 1: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; HR of Bevacizumab Plus Capecitabine vs. Bevacizumab plus Paclitaxel for PFS (stratified) Based on Cox proportional hazards model adjusted by stratification factors at randomization: 1. estrogen and/or progesterone status (positive vs. other) 2. country 3. menopausal status (premenopausal or male <=50 years of age vs. postmenopausal or male >50 years of age); Test type: Superiority — HR is the hazard rate of Bevacizumab Plus Capecitabine divided by hazard rate of Bevacizumab plus Paclitaxel; p = 0.0066, Log Rank; Two-sided log-rank test adjusted by stratification factors at randomization; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [1.08 to 1.61] — HR is the hazard rate of Bevacizumab Plus Capecitabine divided by hazard rate of Bevacizumab plus Paclitaxel

13. Secondary Outcome: Progression Free Survival (PP Population)
Description: as for outcome 12
Time Frame: as for outcome 12
Population: PP population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab Plus Paclitaxel | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 266 | 265
months | 10.9 [10.3 to 12.9] | 8.2 [7.1 to 9.2]
Statistical Analysis 1: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; [analysis description as in outcome 12, analysis 1]; Test type: Superiority — HR is the hazard rate of Bevacizumab plus Capecitabine divided by hazard rate of Bevacizumab plus Paclitaxel; p = 0.0094, Log Rank; Two-sided log-rank test adjusted by stratification factors at randomization; Hazard Ratio (HR) = 1.31, 95% CI 2-sided [1.07 to 1.61] — HR is the hazard rate of Bevacizumab plus Capecitabine divided by hazard rate of Bevacizumab plus Paclitaxel

14. Secondary Outcome: Time to Treatment Failure (ITT Population)
Description: Time to treatment failure (TTF) was defined as time from first drug intake to progression, death or withdrawal from study treatment, whichever occurred first. Patients without an event were censored at the date of the last tumor assessment or last treatment administration, whichever occurred last. Median TTF, associated stratified Hazard Ratio (HR).
Time Frame: From first drug intake to progression, death or withdrawal from study treatment or study closure (whichever occurred first), assessed up to approximately 4.5 years
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab Plus Paclitaxel | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 285 | 279
months | 8.4 [8.0 to 9.7] | 7.2 [6.0 to 8.1]
Statistical Analysis 1: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; HR of Bevacizumab plus Capecitabine vs. Bevacizumab plus Paclitaxel for TTF (stratified) Based on Cox proportional hazards model adjusted by stratification factors at randomization: 1. estrogen and/or progesterone status (positive vs. other) 2. country 3. menopausal status (premenopausal or male <=50 years of age vs. postmenopausal or male >50 years of age); Test type: Superiority — HR is the hazard rate of Bevacizumab plus Capecitabine divided by hazard rate of Bevacizumab plus Paclitaxel; p = 0.1957, Log Rank — Two-sided log-rank test adjusted by stratification factors at randomization; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.94 to 1.35] — HR is the hazard rate of Bevacizumab plus Capecitabine divided by hazard rate of Bevacizumab plus Paclitaxel

15. Secondary Outcome: Time to Treatment Failure (PP Population)
Description: as for outcome 14
Time Frame: as for outcome 14
Population: PP population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab Plus Paclitaxel | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 266 | 265
months | 8.3 [8.0 to 9.4] | 7.3 [5.9 to 8.2]
Statistical Analysis 1: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; [analysis description as in outcome 14, analysis 1]; Test type: Superiority — HR is the hazard rate of Bevacizumab plus Capecitabine divided by hazard rate of Bevacizumab plus Paclitaxel; p = 0.2583, Log Rank — Two-sided log-rank test adjusted by stratification factors at randomization; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.92 to 1.34] — HR is the hazard rate of Bevacizumab plus Capecitabine divided by hazard rate of Bevacizumab plus Paclitaxel

16. Secondary Outcome: Time to Response (ITT Population)
Description: Time to response (TR) was defined as time from randomization until occurrence of response (complete response (CR) or partial response (PR)) according to RECIST criteria. Patients without response were censored after the longest time to response observed in any patient. Median TR, associated stratified Hazard Ratio (HR). Since the median TR was not observed, the number of subjects with a response at given timepoints were reported.
Time Frame: Time from randomization until occurrence of response, assessed up 1.7 years
Population: ITT population, median not reached
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab Plus Paclitaxel | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 285 | 279
Participants
  Month 3 | 83 | 57
  Month 6 | 111 | 69
  Month 9 | 121 | 74
  Month 12 | 123 | 75
  Month 15 | 123 | 75
Statistical Analysis 1: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; HR of Bevacizumab Plus Capecitabine vs. Bevacizumab plus Paclitaxel for TR (stratified) Based on Cox proportional hazards model adjusted by stratification factors at randomization: 1. estrogen and/or progesterone status (positive vs. other) 2. country 3. menopausal status (premenopausal or male <=50 years of age vs. postmenopausal or male >50 years of age); Test type: Superiority — HR is the hazard rate of Bevacizumab Plus Capecitabine divided by hazard rate of Bevacizumab plus Paclitaxel; p = 0.0001, Log Rank — Two-sided log-rank test adjusted by stratification factors at randomization; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.43 to 0.77] — HR is the hazard rate of Bevacizumab Plus Capecitabine divided by hazard rate of Bevacizumab plus Paclitaxel

17. Secondary Outcome: Time to Response (PP Population)
Description: as for outcome 16
Time Frame: Time from randomization until occurrence of response, assessed up 1.7 years
Population: PP population, median not reached
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab Plus Paclitaxel | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 266 | 265
Participants
  Month 3 | 81 | 56
  Month 6 | 108 | 68
  Month 9 | 118 | 72
  Month 12 | 119 | 73
  Month 15 | 119 | 73
Statistical Analysis 1: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; [analysis description as in outcome 16, analysis 1]; Test type: Superiority — HR is the hazard rate of Bevacizumab Plus Capecitabine divided by hazard rate of Bevacizumab plus Paclitaxel; p = 0.0001, Log Rank — Two-sided log-rank test adjusted by stratification factors at randomization; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.41 to 0.75] — HR is the hazard rate of Bevacizumab Plus Capecitabine divided by hazard rate of Bevacizumab plus Paclitaxel

18. Secondary Outcome: Duration of Response (ITT Population)
Description: Duration of response (DR) was defined as time from date of first occurrence of any response (complete response (CR) or partial response (PR)) until the occurrence of progression of disease or death. Patients with response who neither progressed nor died were censored at the date of their last tumor assessment. Median DR, associated stratified Hazard Ratio (HR).
Time Frame: Time from first occurrence of CR or PR until disease progression, death or study closure, whichever occurred first, assessed up to 3.4 years after occurrence of response.
Population: ITT population restricted to patients who experienced a partial or complete response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab Plus Paclitaxel | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 125 | 76
months | 11.2 [10.1 to 14.0] | 10.3 [8.6 to 12.4]
Statistical Analysis 1: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; HR of Bevacizumab Plus Capecitabine vs. Bevacizumab plus Paclitaxel for DR (stratified) Based on Cox proportional hazards model adjusted by stratification factors at randomization: 1. estrogen and/or progesterone status (positive vs. other) 2. country 3. menopausal status (premenopausal or male <=50 years of age vs. postmenopausal or male >50 years of age); Test type: Superiority — HR is the hazard rate of Bevacizumab Plus Capecitabine divided by hazard rate of Bevacizumab plus Paclitaxel; p = 0.0582, Log Rank — Two-sided log-rank test adjusted by stratification factors at randomization; Hazard Ratio (HR) = 1.41, 95% CI 2-sided [0.99 to 2.02] — HR is the hazard rate of Bevacizumab Plus Capecitabine divided by hazard rate of Bevacizumab plus Paclitaxel

19. Secondary Outcome: Duration of Response (PP Population)
Description: as for outcome 18
Time Frame: as for outcome 18
Population: PP population restricted to patients who experienced a partial or complete response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab Plus Paclitaxel | Bevacizumab Plus Capecitabine
Number analyzed (Participants) | 121 | 74
months | 11.2 [9.5 to 14.2] | 10.3 [8.4 to 12.4]
Statistical Analysis 1: Comparison: Bevacizumab Plus Paclitaxel vs Bevacizumab Plus Capecitabine; HR of Arm B vs. Arm A for DR (stratified) Based on Cox proportional hazards model adjusted by stratification factors at randomization: 1. estrogen and/or progesterone status (positive vs. other) 2. country 3. menopausal status (premenopausal or male <=50 years of age vs. postmenopausal or male >50 years of age); Test type: Superiority — HR is the hazard rate of Arm B divided by hazard rate of Arm A; p = 0.0429, Log Rank — Two-sided log-rank test adjusted by stratification factors at randomization; Hazard Ratio (HR) = 1.45, 95% CI 2-sided [1.01 to 2.10] — HR is the hazard rate of Arm B divided by hazard rate of Arm A

ADVERSE EVENTS:
Time Frame: From start of study drug administration until 28 days after the last dose of study medication, assessed up to approximately 5 years
Description: The safety population comprised all patients randomized who received at least one dose of study medication. For the purpose of safety analyses, patients were included in the treatment groups of the treatment actually received. However, if patients received only one component of the assigned combination treatment (e.g. only paclitaxel in group A), then they were analyzed under the Treatment group randomized.
  1 patient in Arm A and 2 patients in Arm B were not treated.
Arm/Group | Bevacizumab Plus Paclitaxel | Bevacizumab Plus Capecitabine
All-Cause Mortality (participants affected / at risk) | 196/284 | 209/277
Serious Adverse Events (participants affected / at risk) | 65/284 | 68/277
Other Adverse Events (participants affected / at risk) | 264/284 | 240/277
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab Plus Paclitaxel (N=284) | Bevacizumab Plus Capecitabine (N=277)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 3 (3) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (4) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain hypoxia (Nervous system disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Nerve root compression (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination, olfactory (Psychiatric disorders) | 1 (1) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Breast lump removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Catheterisation venous (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 2 (2) | 1 (1)
Aortic thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 5 (5)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab Plus Paclitaxel (N=284) | Bevacizumab Plus Capecitabine (N=277)
Anaemia (Blood and lymphatic system disorders) | 35 (59) | 17 (20)
Leukopenia (Blood and lymphatic system disorders) | 46 (127) | 6 (8)
Neutropenia (Blood and lymphatic system disorders) | 87 (204) | 13 (24)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (12) | 19 (26)
Abdominal pain (Gastrointestinal disorders) | 20 (26) | 18 (21)
Abdominal pain upper (Gastrointestinal disorders) | 18 (24) | 14 (17)
Constipation (Gastrointestinal disorders) | 27 (32) | 25 (32)
Diarrhoea (Gastrointestinal disorders) | 58 (83) | 59 (83)
Dyspepsia (Gastrointestinal disorders) | 17 (24) | 15 (17)
Nausea (Gastrointestinal disorders) | 57 (82) | 70 (94)
Stomatitis (Gastrointestinal disorders) | 22 (27) | 20 (24)
Vomiting (Gastrointestinal disorders) | 29 (40) | 34 (46)
Asthenia (General disorders) | 44 (50) | 34 (37)
Fatigue (General disorders) | 97 (127) | 76 (89)
Mucosal inflammation (General disorders) | 23 (29) | 13 (13)
Oedema peripheral (General disorders) | 27 (28) | 11 (13)
Pyrexia (General disorders) | 23 (27) | 17 (20)
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 (3) | 16 (18)
Urinary tract infection (Infections and infestations) | 24 (29) | 14 (18)
Decreased appetite (Metabolism and nutrition disorders) | 35 (38) | 33 (38)
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 (58) | 18 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 27 (35) | 29 (29)
Bone pain (Musculoskeletal and connective tissue disorders) | 28 (33) | 29 (31)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 14 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 20 (26) | 9 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 (32) | 24 (28)
Dizziness (Nervous system disorders) | 33 (39) | 17 (19)
Dysgeusia (Nervous system disorders) | 17 (19) | 10 (14)
Headache (Nervous system disorders) | 37 (46) | 27 (32)
Neuropathy peripheral (Nervous system disorders) | 86 (105) | 9 (9)
Paraesthesia (Nervous system disorders) | 17 (18) | 12 (12)
Peripheral sensory neuropathy (Nervous system disorders) | 23 (25) | 5 (5)
Polyneuropathy (Nervous system disorders) | 27 (35) | 6 (7)
Proteinuria (Renal and urinary disorders) | 10 (13) | 16 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 32 (37) | 20 (22)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 35 (37) | 10 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 32 (39) | 24 (27)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 89 (122) | 39 (46)
Alopecia (Skin and subcutaneous tissue disorders) | 87 (88) | 5 (5)
Nail disorder (Skin and subcutaneous tissue disorders) | 48 (50) | 10 (10)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 8 (8) | 155 (197)
Rash (Skin and subcutaneous tissue disorders) | 17 (20) | 11 (14)
Hypertension (Vascular disorders) | 102 (192) | 83 (130)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes